CLINICAL TRIAL: NCT05079984
Title: Agile Development of a Digital Exposure Treatment for Youth With Chronic Musculoskeletal Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Karolinska Institutet (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Lauren Harrison, Clinical Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 53323; 1K23AR079608-01 (NIH)
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Exposure; Adolescent Behavior; Child Behavior
MeSH Terms: conditions — Chronic Pain; Adolescent Behavior; Child Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Graded Exposure Intervention (Experimental): For Aim 2, adolescents with chronic pain will be enrolled in a single-arm feasibility trial examining acceptability, feasibility, and preliminary effectiveness of a novel, digitally delivered, graded exposure treatment.
  Interventions: Behavioral: Graded exposure treatment (GET)

INTERVENTIONS:
Behavioral: Graded exposure treatment (GET) — Graded-exposure is a theory driven, individually tailored, and evidenced based behavioral intervention for individuals with chronic pain targeting pain-related impairment by exposing patients to previously feared and avoided activities.

SUMMARY:
This project proposes to systematically develop and evaluate the feasibility and preliminary effectiveness of a digitally delivered, graded exposure treatment for youth with chronic musculoskeletal pain, utilizing a sequential replicated and randomized single-case experimental design (SCED). SCED provides the opportunity to rigorously evaluate treatment effectiveness at the individual level.

Development of iGET Living will be based on a series of short iterations, with alpha testing (Aim 1) on a small sample of adolescents with chronic pain (N = 15). For Aim 1, participants will participate in three, two hour focus groups (one per week over the course of three weeks), resulting in 6 total hours of participation per participant for Aim 1.

Aim 2 will involve a sample (N = 20 youth) of naïve end-users. Participants will be enrolled in a baseline period ranging from 7-25 days (done to support SCED methodology) after which they will be enrolled in the online intervention program, lasting 6-weeks. Patients will be contacted 3-months post-discharge from treatment (week 22 of enrollment) and will complete self-report outcome measures at this time.

ELIGIBILITY:
Inclusion Criteria:

* Youth ages 10-18
* Have diagnosis of chronic musculoskeletal pain (>3months)
* Have moderate to high pain interference (PROMIS Pain Interference ≥ 61)
* English literate
* Have access to computer, smartphone, or tablet with internet connection

Exclusion Criteria:

* Significant cognitive impairment (e.g., brain injury)
* Significant medical or psychiatric problems that would interfere with treatment

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Acceptability of Treatment Content and Digital Delivery Questionnaire - Likert Scale (Aim 1 and Aim 2) | Baseline through 3-month follow-up (up to 22 weeks)
  Participant-rated acceptability measured on 5-point Likert scale. Range 0-4 (higher scores indicate more acceptable). Questionnaire will be administered to youth with chronic pain and their parents.
Assessment of Acceptability of Treatment Content and Digital Delivery Questionnaire - Participant Responses (Aim 1 and Aim 2) | Baseline through 3-month follow-up (up to 22 weeks)
  Acceptability will be assessed qualitatively through participant responses to open-ended questions related to acceptability, ease of use, comprehensibility, and suggestions for improvement. Responses will be assessed categorically by the investigator. Questionnaire will be administered to youth with chronic pain and their parents.
Participant Satisfaction with the Intervention (Aim 1 and Aim 2) | 19 weeks (Assessed at the end of treatment)
  Treatment satisfaction at the end of treatment will be evaluated by examining mean satisfaction scores on an adapted version of the Pain Service Satisfaction Test (PSST, McCracken et al., 1997). The PSST consists of 23 items rated on a 5-point Likert Scale (0 = not at all satisfied to 4 = very satisfied) and assesses the patient and parent's experience of the intervention. Scores range from 0-92. A score greater than/equal to 40 of 60 (satisfied to very satisfied) will indicate high levels of satisfaction with the intervention content.
Percentage of Participants Dropped Out of Intervention (Aim 2) | 19 weeks (Assessed at the end of treatment)
  As a measure of treatment adherence, we will calculate the percentage of participants who drop out or withdraw from the intervention prior to completion of the intervention.
Expectations for Treatment (Aim 2) | Baseline (up to 2 minutes to complete the survey)
  Participants (child) and parent expectations for treatment will be measured by the Treatment Expectancy and Creditability, Borkovec & Nau, 1972). The TEC is comprised of 6 items rated on a 0 to 10 Likert-scale assessing expectations related to the effectiveness of the current treatment. The TEC is completed by the patient at the end of the first treatment session. Higher scores indicate greater expectations for treatment effectiveness.
Functional Disability (Aim 2) | Baseline through 3-month follow-up (up to 22 weeks)
  Functional disability will be assessed using the Functional Disability Inventory (FDI, Walker & Greene, 1991), a 15-item self-report measure of perceived difficulty in performing activities in school, home, physical, and social contexts. Items are rated on a 5-point Likert scale ranging from 0 (no trouble) to 4 (impossible). Items are summed to create a total score (range 0-60), with higher scores indicating greater disability.

SECONDARY OUTCOMES:
Child Fear of Pain (Aim 2) | Baseline through 3-month follow-up (up to 22 weeks)
  Fear of Pain Questionnaire- Child (FOPQ-C, Simons et al., 2011) consists of 24 items, with each item rated on a 5-point Likert scale (0 = "strongly disagree" to 4 = "strongly agree"). The FOPQ-C contains two subscales: Fear of Pain (11 items) and Avoidance of Activities (13 items). Total score is derived by summing subscale items, with higher scores indicating greater pain related fear (score range 0-44) and avoidance of activities (score range 0-52).
Parental Fear of Pain (Aim 2) | Baseline through 3-month follow-up (up to 22 weeks)
  The Parent Fear of Pain Questionnaire (PFOPQ, Simons et al., 2015) assesses parent's fear associated with their child's pain experiences. The PFOPQ contains 23 items assessed on a 5-point Likert scale (0 = "strongly disagree" to 4 "strongly agree"). Items are summed to create a total score (0-92), with higher scores indicated greater parent fear associated with their child's pain.
Child Pain Catastrophizing (Aim 2) | Baseline through 3-month follow-up (up to 22 weeks)
  The Pain Catastrophizing Scale -Child Version (PCS-C, Crombez et al., 2003) assesses negative cognitions associated with pain. The PCS-C is comprised of 13-items rated on a 5-point Likert scale (0= "not at all true" to 4 "very true"). A total score (0-52) is obtained by summing all items. Higher scores indicate higher levels of catastrophic thinking.
Parent Pain Catastrophizing (Aim 2) | Baseline through 3-month follow-up (up to 22 weeks)
  Pain Catastrophizing Scale-Parent Version (PCS-P, Goubert et al., 2006) assesses parents' negative cognitions associated with their child's pain. It is comprised of 13 items rated on a 5-point Likert scale (0 = "not true at all" to 4 = "very true"). A total score (0-52) is derived by summing items, with higher scores indicating higher levels of catastrophic thinking.
Child Pain Acceptance (Aim 2) | Baseline through 3-month follow-up (up to 22 weeks)
  Child report on the Chronic Pain Acceptance Questionnaire for Adolescents-short form (CPAQ-A8, Gauntlett-Gilbert et al., 2018) will be used to assess pain acceptance in the child. The CPAQ-A8 is an 8-item measure consisting of two subscales: Activity Engagement (4 items) and Pain Willingness (4 items). Items are rated on a 5-point Likert scale ranging from 0 (Never True) to 4 (Always True) and yield a total score for each subscale ranging from 0-16. Higher scores indicate greater Activity Engagement and greater Pain Willingness .
Parent Psychological Flexibility (Aim 2) | Baseline through 3-month follow-up (up to 22 weeks)
  The Parent Psychological Flexibility Questionnaire (PPFQ-10, Timmers et al., 2019) is a 10-item parent self-report questionnaire assessing a parent's ability to accept their own distress and respond adaptively and flexibly to their child's pain. Items are rated on a 5-point Likert scale (0= " never true" to 4 = "always true") and are summed to create a total score, ranging from 0 - 40. Higher scores indicate greater parent psychological flexibility.
Parent Responses to Childs Pain (Aim 2) | Baseline through 3-month follow-up (up to 22 weeks)
  Adult Responses to Children's Symptoms (ARCS, Claar et al., 2010) assesses parents' behavioral responses to children's pain behaviors. The Protect subscale (13 items) will be utilized in this study. The Protect scale refers to protective parental behavior, such as giving the child special attention and limiting the child's normal activities and responsibilities. All items are rated on a 5-point Likert scale (0 = "never" to 4 "always"), and are averaged to create a total score ranging from 0-4. Hiigher scores indicating greater use of a particular type of response to their child's pain.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E Harrison, PhD, Principal Investigator — Stanford University
Locations (1):
- Pediatric Pain Management Clinic, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huguet A, Miro J. The severity of chronic pediatric pain: an epidemiological study. J Pain. 2008 Mar;9(3):226-36. doi: 10.1016/j.jpain.2007.10.015. Epub 2007 Dec 21. PMID 18088558
- [Background] King S, Chambers CT, Huguet A, MacNevin RC, McGrath PJ, Parker L, MacDonald AJ. The epidemiology of chronic pain in children and adolescents revisited: a systematic review. Pain. 2011 Dec;152(12):2729-2738. doi: 10.1016/j.pain.2011.07.016. PMID 22078064
- [Background] Wilson K, Bell C, Wilson L, Witteman H. Agile research to complement agile development: a proposal for an mHealth research lifecycle. NPJ Digit Med. 2018 Sep 13;1:46. doi: 10.1038/s41746-018-0053-1. eCollection 2018. PMID 31304326
- [Background] Groenewald CB, Essner BS, Wright D, Fesinmeyer MD, Palermo TM. The economic costs of chronic pain among a cohort of treatment-seeking adolescents in the United States. J Pain. 2014 Sep;15(9):925-33. doi: 10.1016/j.jpain.2014.06.002. Epub 2014 Jun 19. PMID 24953887
- [Background] Murray CB, Groenewald CB, de la Vega R, Palermo TM. Long-term impact of adolescent chronic pain on young adult educational, vocational, and social outcomes. Pain. 2020 Feb;161(2):439-445. doi: 10.1097/j.pain.0000000000001732. PMID 31651579
- [Background] Groenewald CB, Patel KV, Rabbitts JA, Palermo TM. Correlates and motivations of prescription opioid use among adolescents 12 to 17 years of age in the United States. Pain. 2020 Apr;161(4):742-748. doi: 10.1097/j.pain.0000000000001775. PMID 31815917
- [Background] Peng P, Stinson JN, Choiniere M, Dion D, Intrater H, Lefort S, Lynch M, Ong M, Rashiq S, Tkachuk G, Veillette Y; STOPPAIN Investigators Group. Dedicated multidisciplinary pain management centres for children in Canada: the current status. Can J Anaesth. 2007 Dec;54(12):985-91. doi: 10.1007/BF03016632. PMID 18056207
- [Background] Eccleston C, Blyth FM, Dear BF, Fisher EA, Keefe FJ, Lynch ME, Palermo TM, Reid MC, Williams ACC. Managing patients with chronic pain during the COVID-19 outbreak: considerations for the rapid introduction of remotely supported (eHealth) pain management services. Pain. 2020 May;161(5):889-893. doi: 10.1097/j.pain.0000000000001885. No abstract available. PMID 32251203
- [Background] Vlaeyen JWS, Linton SJ. Fear-avoidance and its consequences in chronic musculoskeletal pain: a state of the art. Pain. 2000 Apr;85(3):317-332. doi: 10.1016/S0304-3959(99)00242-0. PMID 10781906
- [Background] Vlaeyen JWS, Crombez G, Linton SJ. The fear-avoidance model of pain. Pain. 2016 Aug;157(8):1588-1589. doi: 10.1097/j.pain.0000000000000574. No abstract available. PMID 27428892
- [Background] Vlaeyen JW, de Jong J, Geilen M, Heuts PH, van Breukelen G. The treatment of fear of movement/(re)injury in chronic low back pain: further evidence on the effectiveness of exposure in vivo. Clin J Pain. 2002 Jul-Aug;18(4):251-61. doi: 10.1097/00002508-200207000-00006. PMID 12131067
- [Background] Simons LE, Harrison LE, O'Brien SF, Heirich MS, Loecher N, Boothroyd DB, Vlaeyen JWS, Wicksell RK, Schofield D, Hood KK, Orendurff M, Chan S, Lyons S. Graded exposure treatment for adolescents with chronic pain (GET Living): Protocol for a randomized controlled trial enhanced with single case experimental design. Contemp Clin Trials Commun. 2019 Sep 10;16:100448. doi: 10.1016/j.conctc.2019.100448. eCollection 2019 Dec. PMID 31650069
- [Background] Simons LE, Sieberg CB, Carpino E, Logan D, Berde C. The Fear of Pain Questionnaire (FOPQ): assessment of pain-related fear among children and adolescents with chronic pain. J Pain. 2011 Jun;12(6):677-86. doi: 10.1016/j.jpain.2010.12.008. Epub 2011 Feb 26. PMID 21354866
- [Background] Walker LS, Greene JW. The functional disability inventory: measuring a neglected dimension of child health status. J Pediatr Psychol. 1991 Feb;16(1):39-58. doi: 10.1093/jpepsy/16.1.39. PMID 1826329
- [Background] Simons LE, Smith A, Kaczynski K, Basch M. Living in fear of your child's pain: the Parent Fear of Pain Questionnaire. Pain. 2015 Apr;156(4):694-702. doi: 10.1097/j.pain.0000000000000100. PMID 25630026
- [Background] Goubert L, Eccleston C, Vervoort T, Jordan A, Crombez G. Parental catastrophizing about their child's pain. The parent version of the Pain Catastrophizing Scale (PCS-P): a preliminary validation. Pain. 2006 Aug;123(3):254-263. doi: 10.1016/j.pain.2006.02.035. Epub 2006 Apr 27. PMID 16644128
- [Background] Claar RL, Guite JW, Kaczynski KJ, Logan DE. Factor structure of the Adult Responses to Children's Symptoms: validation in children and adolescents with diverse chronic pain conditions. Clin J Pain. 2010 Jun;26(5):410-7. doi: 10.1097/AJP.0b013e3181cf5706. PMID 20473048
- [Background] Crombez G, Bijttebier P, Eccleston C, Mascagni T, Mertens G, Goubert L, Verstraeten K. The child version of the pain catastrophizing scale (PCS-C): a preliminary validation. Pain. 2003 Aug;104(3):639-646. doi: 10.1016/S0304-3959(03)00121-0. PMID 12927636
- [Background] Timmers I, Simons LE, Hernandez JM, McCracken LM, Wallace DP. Parent psychological flexibility in the context of pediatric pain: Brief assessment and associations with parent behaviour and child functioning. Eur J Pain. 2019 Aug;23(7):1340-1350. doi: 10.1002/ejp.1403. Epub 2019 May 14. PMID 31002473
- [Background] Gauntlett-Gilbert J, Alamire B, Duggan GB. Pain Acceptance in Adolescents: Development of a Short Form of the CPAQ-A. J Pediatr Psychol. 2019 May 1;44(4):453-462. doi: 10.1093/jpepsy/jsy090. PMID 30496433
- [Background] Palermo T. Remote management of pediatric pain. Encyclopedia of Pain 2nd Edition New York: Springer 2013:3389-93
- [Background] Borkovec TD, & Nau, S. D. . Credibility of analogue therapy rationales. Journal of Behavior Therapy and Experimental Psychology 1972;3:257-60
- [Background] Simons LE, Vlaeyen JWS, Declercq L, Smith AM, Beebe J, Hogan M, Li E, Kronman CA, Mahmud F, Corey JR, Sieberg CB, Ploski C. Avoid or engage? Outcomes of graded exposure in youth with chronic pain using a sequential replicated single-case randomized design. Pain. 2020 Mar;161(3):520-531. doi: 10.1097/j.pain.0000000000001735. PMID 31693541
- [Background] McCracken LM, Klock PA, Mingay DJ, Asbury JK, Sinclair DM. Assessment of satisfaction with treatment for chronic pain. J Pain Symptom Manage. 1997 Nov;14(5):292-9. doi: 10.1016/s0885-3924(97)00225-x. PMID 9392923
- [Derived] Harrison LE, Webster SN, Van Orden AR, Choate E, Jehl N, Stinson J, Wicksell RK, Bonnert M, Lalouni M, Darnall BD, Simons LE. Agile development of a digital exposure treatment for youth with chronic musculoskeletal pain: protocol of a user-centred design approach and examination of feasibility and preliminary efficacy. BMJ Open. 2022 Sep 15;12(9):e065997. doi: 10.1136/bmjopen-2022-065997. PMID 36109029